CLINICAL TRIAL: NCT00314028
Title: Promoting HIV Risk Reduction Among African American Men
Brief Title: Effectiveness of HIV Risk Reduction Program Among African American Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Richard Crosby (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Richard Crosby, PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21MH066682 (NIH); R21MH066682 (NIH); DAHBR 9A-ASPQ
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Sexually Transmitted Diseases; HIV
Keywords: African American; Men; Sexually Transmitted Diseases; Condoms
MeSH Terms: conditions — Sexually Transmitted Diseases; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Active Comparator): Standard of care treatment
  Interventions: Other: Control standard of care treatment
- 2 (Experimental): Educational program designed to motivate and provide information on the correct use of condoms
  Interventions: Behavioral: Focus on the Future; Other: Control standard of care treatment

INTERVENTIONS:
Behavioral: Focus on the Future — Focus on the Future is an educational program designed to promote proper condom use.
  Arms: 2
Other: Control standard of care treatment — Standard of care treatment is the normal treatment that someone would receive for the particular sexually transmitted disease or virus.

SUMMARY:
This study will test the effectiveness of a brief clinic-based program designed to promote the correct use of condoms among young African-American men newly diagnosed with a sexually transmitted disease.

DETAILED DESCRIPTION:
Sexually transmitted diseases (STDs), including HIV infections, are most commonly spread through unprotected sexual intercourse. STDs are a major health concern, especially among young ethnic minorities in the United States. The rate of STDs is significantly greater in urban areas where ethnic minorities, particularly African-American males, are commonly represented. Despite this knowledge, safe sexual practices, including correct condom use, are not the norm among minority males. It is believed that educational outreach designed to motivate and inform on the correct use of condoms will be effective in encouraging safer sex practices. This study will test the effectiveness of a brief clinic-based program designed to promote the correct use of condoms among young African-American men newly diagnosed with an STD.

Participants in this single blind study will be randomly assigned to an experimental or control group. Upon being diagnosed with an STD, men in both groups will receive standard of care follow-up treatment. Men in the experimental group will also receive a one-on-one educational session on condom use. The educational session will be led by a health educator and will last about 30 minutes, depending on the existing skills and learning abilities of the participants. Using information provided by the participants on past experience with condoms, the health educator will attempt to correct misunderstandings about and problems with condom use. Upon enrollment, all men will respond to a series of pre-recorded questions and will be required to demonstrate their ability to apply condoms to a penile model. The same questions and procedure will be repeated 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as African American
* Clinically diagnosed with an STD
* Reports at least one episode of condom use with a female within 3 months of study entry (this requirement does not restrict men who also have sex with men from study participation)
* Fluent in English

Exclusion Criteria:

* Known HIV infection

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2003-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Frequency of unprotected penile vaginal sex | Measured at Month 3

SECONDARY OUTCOMES:
Frequency of condom use errors and problems | Measured at Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Forsythe, PhD, Study Chair — National Institute of Mental Health (NIMH)